CLINICAL TRIAL: NCT03079219
Title: A Randomized Study to Determine the Efficacy and Tolerability of Olanzapine for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Chinese Breast Cancer Patients
Brief Title: Olanzapine for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Chinese Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CCTU (Other)
Responsible Party: Sponsor-Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYM010
Record Dates: First submitted 2017-02-08; First posted 2017-03-14 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Aprepitant, Ondansetron, Dexamethasone and Olanzapine
  Interventions: Drug: Experimental drug: Aprepitant; Drug: Experimental drug: Ondansetron; Drug: Experimental drug: Dexamethasone; Drug: Experimental drug: Olanzapine
- Standard (Other): Aprepitant, Ondansetron, Dexamethasone
  Interventions: Drug: Standard: Aprepitant; Drug: Standard: Ondansetron; Drug: Standard: Dexamethasone

INTERVENTIONS:
Drug: Experimental drug: Aprepitant — Day 1: 125mg QD; Day 2 to Day 3: 80mg QD
  Arms: Experimental
Drug: Experimental drug: Ondansetron — Day 1: 8mg BD, First dose 8mg, Second dose 8mg, 8 hours after first dose
  Arms: Experimental
Drug: Experimental drug: Dexamethasone — Day 1: 12mg QD
  Arms: Experimental
Drug: Experimental drug: Olanzapine — Day 1 to Day 5: 10mg QD
  Arms: Experimental
Drug: Standard: Aprepitant — Day 1: 125mg QD, Day 2 to Day3: 80mg QD
  Arms: Standard
Drug: Standard: Ondansetron — Day 1: 8mg BD, First dose 8mg, second dose 8mg, 8 hours after first dose
  Arms: Standard
Drug: Standard: Dexamethasone — Day 1: 12mg QD ; Day 2 to Day 3: 4mg BD
  Arms: Standard

SUMMARY:
The Olanzapine Regimen will be superior to the Standard Regimen, as measured by the proportion of patients with Complete Response in the 120 hours following AC chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Chinese patient, female >=18 and < 75 years of age.
* Patient is diagnosed with early breast cancer.
* Patient is naïve to emetogenic chemotherapy moderately or highly emetogenecity.
* Patient is scheduled to receive her first course of adjuvant chemotherapy for breast cancer follows:
* IV adriamycin 60 mg/m2 + cyclophosphamide 600 mg/m2
* Patient has a predicted life expectancy of >=4 months.
* Patient has ECOG Performance Status of 0-1
* Premenopausal female patients must not be pregnant (documented negative urine pregnancy test).
* Patient is able to read, understand and complete study questionnaires and diary, including questions requiring a visual analog scale (VAS) response.
* Patient understands the procedures and agrees to participate in the study by giving written informed consent

Exclusion Criteria:

* Patient with advanced breast cancer.
* Patient receiving cisplatin or any other chemotherapy of higher emetogenic potential, except for cyclophosphamide and doxorubicin in the regimens described above.
* Patients who are scheduled to receive concurrent radiation as part of their chemotherapy regimen for their malignancy
* Patients who experience any vomiting or grade 2-3 nausea per Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v 4.03) in the 24 hours before Day 1 of chemotherapy
* Patient has a history of treatment with moderately to highly emetogenic chemotherapy.
* Patient has an active infection (e.g., pneumonia, systemic fungal infection) or any uncontrolled disease (e.g., diabetes mellitus, hypertension) which, in the opinion of the investigator, might confound the results of the study or pose unwarranted risk.
* Patient with history of glaucoma, dementia, seizures, Parkinson's disease, Neuroleptic Malignant Syndrome (NMS), thromboembolic events.
* Patient currently uses any illicit drugs, including marijuana, or has current evidence of alcohol abuse as determined by the investigator.
* Patient is mentally incapacitated or has a significant emotional or psychiatric disorder that, in the opinion of the investigator, precludes study entry.
* Patients who are regular alcohol drinker or smoker
* Patient has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose unwarranted risk.
* Patient has a history of hypersensitivity to aprepitant, ondansetron or dexamethasone.
* Patients who have phenylketonuria and abnormal uric acid.
* Any investigational drugs taken within 4 weeks prior to Day 1 of cycle 1, and/or is scheduled to receive any investigational drug during the study;
* Patient is taking systemic corticosteroid therapy at any dose; however, topical and inhaled corticosteroids are permitted.
* Patient has taken a non-registered investigational drug within the 28 days of the Prestudy Visit.
* Use, in the 28 days prior to Treatment Day 1, of barbiturates, rifampicin or rifabutin, phenytoin or carbamazepine
* Use, in the 7 days prior to Treatment Day 1, of terfenadine, cisapride, astemizole, clarithromycin (azithromycin, erythromycin and roxithromycin are permitted), ketoconazole or itraconazole (fluconazole is permitted), amifostine pimozide 5-HT3 antagonists (ondansetron, granisetron, dolasetron, or tropisetron) phenothiazines (e.g., prochlorperazine, fluphenazine, perphenazine, thiethylperazine, or chlorpromazine) butyrophenones (e.g., haloperidol or droperidol) benzamides (e.g., metoclopramide or alizapride) domperidone cannabinoids NK1 receptor antagonists
* Use, in the 48 hours prior to Treatment Day 1, of benzodiazepines or opiates, except for single daily doses of lorazepam.

  s. Use of the following drugs: carbamazepine Fluvoxamine ciprofloxacin dopamine agonists. antiparkinsonian medicinal products medicinal products known to increase QTc interval t. Abnormal laboratory values

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Number of episodes of nausea in the first 120 hours after first cycle of chemotherapy. | 120 hours
  Number of episodes of nausea in the first 120 hours after first cycle of chemotherapy.
Number of episodes of vomiting in the first 120 hours after first cycle of chemotherapy. | 120 hours
  Number of episodes of vomiting in the first 120 hours after first cycle of chemotherapy.

SECONDARY OUTCOMES:
Number of episodes of nausea in the first 120 hours during 4 cycles of chemotherapy. | 120 hours
  Number of episodes of nausea in the first 120 hours during 4 cycles of chemotherapy.
Number of episodes of vomiting in the first 120 hours during 4 cycles of chemotherapy. | 120 hours
  Number of episodes of vomiting in the first 120 hours during 4 cycles of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Yeo, MD, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided